CLINICAL TRIAL: NCT02108925
Title: Oxygen Supply and Ventilation During Physical Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Oxygen Supplementation During Exercise in Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/2396
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypoxia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supplementary oxygen (Experimental): Study subjects receive, in randomized order, either supplementary 30% oxygen or air (21% Oxygen) from a gas tight bag
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — supplementary oxygen during exercise

SUMMARY:
The project will test the hypothesis that lung ventilation during exercise is unaffected by oxygen supplementation. In addition, the acute effect of oxygen supplementation on dyspnoea, heart rate and blood pressure will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease

Exclusion Criteria:

* No exacerbation
* No active heart disease

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary ventilation | 1 hour

SECONDARY OUTCOMES:
Dyspnoea | 1 hour
Heart rate | 1 hour
Blood pressure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anne Edvardsen, PhD, Principal Investigator — LHL Helse
Locations (1):
- LHL-klinikkene Glittre, Hakadal, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No